CLINICAL TRIAL: NCT00184431
Title: A Randomized Controlled Trial Comparing Intensive Task Specific Training With Traditional Follow up Care After Discharge From a Stroke Unit.
Brief Title: Does Intensive Task Specific Training Improve Balance After Acute Stroke?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU01-ISM-NTNU
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Cerebrovascular Accident
Keywords: Cerebrovascular Accident; Physical Therapy Techniques; Musculoskeletal Equilibrium; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Intensive task specific balance training
  Interventions: Behavioral: Physical therapy technique and exercises
- B (Active Comparator): Traditional physical therapy
  Interventions: Behavioral: Physical therapy technique and exercises

INTERVENTIONS:
Behavioral: Physical therapy technique and exercises — The experimental group receives task specific physical therapy three times a week for the first four weeks after discharge from hospital and one session pr week for the next eight weeks in addition to ordinary physical therapy The active comparator group receives only ordinary physical therapy during this period.

SUMMARY:
The aim of this study is to investigate whether additional task specific physiotherapy treatment and a self administrated home training program results in better balance compared to traditional follow up care.

DETAILED DESCRIPTION:
Increased risk of falling is a major problem after stroke and impaired balance is one of the main reasons for falling. Early and intensive physiotherapy seems to be beneficial for functional outcome after stroke although it is still unknown whether one specific physiotherapy technique is better than another.

Comparison: Traditional follow up care by the community health care system with additional task specific physiotherapy three times a week and a daily self administrated home training program compared to traditional follow up care by the community health care system.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the stroke unit with a diagnosis of stroke
* Living in the city of Trondheim
* Included 4 - 14 days after first sign of symptoms
* Modified Rankin Scale > 3 before admission to hospital
* Scandinavian Stroke Scale (SSS) less than 58 points and more than 14 points
* SSS leg item less than 6 points or SSS movement item less than 12 points
* Discharged to home or a rehabilitation clinic
* Mini Mental State Examination Score more than 20 points
* Able and willing to provide informed consent

Exclusion Criteria:

* Seriously heart- and lung-diseases
* Other diseases which makes it difficult to evaluate the function
* Already included in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The Berg Balance Scale | Inclusion, four weeks follow-up, twelve weeks follow-up and six months follow-up

SECONDARY OUTCOMES:
Mini Mental State Examination | Inclusion
Scandinavian Stroke Scale | Inclusion
Motor Assessment Scale | Inclusion, four weeks follow-up, twelve weeks follow-up, six months follow-up
Timed Up and Go | Inclusion, four weeks follow-up, twelve weeks follow-up, six months follow-up
Step Test | Inclusion, four weeks follow-up, twelve weeks follow-up, six months follow-up
Walking speed | Inclusion, four weeks follow-up, twelve weeks follow-up, six months follow-up
Barthel Index | Inclusion, four weeks follow-up, twelve weeks follow-up, six months follow-up
Modified Rankin Scale | Inclusion, four weeks follow-up, twelve weeks follow-up, six months follow-up
Fall Efficacy Scale | Inclusion, four weeks follow-up, twelve weeks follow-up, six months follow-up
Stroke Impact Scale | Inclusion, four weeks follow-up, twelve weeks follow-up, six months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bent Indredavik, assoc-prof, Study Chair — Department of Neuroscience, Faculty of Medicine, Norwegian university of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Askim T, Morkved S, Engen A, Roos K, Aas T, Indredavik B. Effects of a community-based intensive motor training program combined with early supported discharge after treatment in a comprehensive stroke unit: a randomized, controlled trial. Stroke. 2010 Aug;41(8):1697-703. doi: 10.1161/STROKEAHA.110.584284. Epub 2010 Jun 17. PMID 20558830